CLINICAL TRIAL: NCT05173987
Title: A Phase 3 Randomized, Open-label, Active-comparator Controlled Clinical Study of Pembrolizumab Versus Platinum Doublet Chemotherapy in Participants With Mismatch Repair Deficient (dMMR) Advanced or Recurrent Endometrial Carcinoma in the First-line Setting (KEYNOTE-C93/GOG-3064/ENGOT-en15)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Chemotherapy in Mismatch Repair Deficient (dMMR) Advanced or Recurrent Endometrial Carcinoma (MK-3475-C93/KEYNOTE-C93/GOG-3064/ENGOT-en15)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-C93; MK-3475-C93 (Other: MSD); KEYNOTE-C93 (Other: MSD); GOG-3064 (Other: Gynecologic Oncology Group (GOG)); ENGOT-en15 (Other: European Network of Gynaecological Oncological Trial Groups (ENGOT)); jRCT2011210065 (Registry Identifier: jRCT); 2021-003185-12 (EudraCT Number)
Record Dates: First submitted 2021-12-20; First posted 2021-12-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 400 mg via IV infusion on Day 1 of each 6-week cycle (Q6W) for up to 18 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab
- Carboplatin+paclitaxel (Active Comparator): Participants receive a combination of paclitaxel 175 mg/m^2 on Day 1 of each 3-week cycle (Q3W) and carboplatin AUC 5 or 6 on Day 1 Q3W for 6 cycles (up to approximately 4 months). Participants who experience a severe hypersensitivity reaction to paclitaxel or an adverse event (AE) requiring discontinuation of paclitaxel may receive docetaxel 75 mg/m^2 in place of paclitaxel on Day 1 Q3W after Sponsor consultation. Participants who experience a severe hypersensitivity reaction to carboplatin or an AE requiring discontinuation of carboplatin may receive cisplatin 75 mg/m^2 in place of carboplatin on Day 1 Q3W after Sponsor consultation.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: docetaxel; Drug: cisplatin

INTERVENTIONS:
Biological: pembrolizumab — Intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: carboplatin — IV infusion
  Other Names: PARAPLATIN®
  Arms: Carboplatin+paclitaxel
Drug: paclitaxel — IV infusion
  Other Names: TAXOL®
  Arms: Carboplatin+paclitaxel
Drug: docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Carboplatin+paclitaxel
Drug: cisplatin — IV infusion
  Other Names: PLATINOL-AQ®
  Arms: Carboplatin+paclitaxel

SUMMARY:
The purpose of this study is to assess the safety and efficacy of treatment with pembrolizumab (MK-3475) compared to a combination of carboplatin and paclitaxel in women with mismatch repair deficient (dMMR) advanced or recurrent endometrial carcinoma who have not previously been treated with prior systemic chemotherapy.

The primary study hypotheses are that pembrolizumab is superior to the combination of carboplatin and paclitaxel with respect to Progression Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) and Overall Survival (OS).

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a histologically confirmed diagnosis of inoperable, Stage III or IV or recurrent Endometrial Carcinoma (EC) or carcinosarcoma (mixed Mullerian tumor) that is centrally confirmed as dMMR.
* Has radiographically evaluable disease, either measurable or non-measurable per RECIST 1.1, as assessed by the investigator. Note: primary Stage IVB that has undergone surgical resection is allowed regardless of presence of measurable or evaluable disease.
* Has received no prior systemic therapy for EC except for the following:

  1. May have received 1 prior line of systemic platinum-based adjuvant and/or neoadjuvant chemotherapy in the setting of curative-intent resection if the recurrence occurred ≥6 months after the last dose of chemotherapy.
  2. May have received prior radiation with or without radiosensitizing chemotherapy if >2 weeks before the start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
  3. May have received prior hormonal therapy for treatment of EC, provided that it was discontinued ≥1 week prior to randomization.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before randomization.
* Is not pregnant or breastfeeding and agrees to not donate eggs and use a highly effective contraceptive method for 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapy if a woman of childbearing potential (WOCBP).
* Has a negative highly sensitive pregnancy test (urine or serum) within 24 hours for urine or 72 hours for serum before the first dose of study intervention if a WOCBP.
* Provides an archival tumor tissue sample or newly obtained (core, incisional, or excisional) biopsy of a tumor lesion not previously irradiated for verification of dMMR status and histology.
* If Hepatitis B surface antigen (HBsAg) positive, has received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and has undetectable HBV viral load prior to randomization.
* If has a history of Hepatitis C virus (HCV) infection, has undetectable HCV viral load at screening.

Exclusion Criteria:

* Has uterine mesenchymal tumor such as an endometrial stromal sarcoma, leiomyosarcoma, or other types of pure sarcomas. Adenosarcomas and neuroendocrine tumors are not allowed.
* Has EC of any histology that is proficient mismatch repair (pMMR).
* Is a candidate for curative-intent surgery or curative-intent radiotherapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], Tumor necrosis factor receptor superfamily, member 4 [OX 40], tumor necrosis factor receptor superfamily member 9 [CD137]).
* Has received prior systemic anticancer therapy including investigational agents for any advanced or metastatic EC. (Note: Prior chemotherapy administered as adjuvant therapy, neoadjuvant therapy, and/or concurrently with radiation is permitted.
* Has had a major operation and has not recovered adequately from the procedure and/or any complications from the operation before starting study intervention.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Is currently participating in or has participated in a study of an investigational agent for EC, has participated in a study of an investigational agent for non-EC within 4 weeks before the first dose of study intervention, or has used an investigational device within 4 weeks before the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (excluding carcinoma in situ of the bladder) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has a known intolerance to any study intervention and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection, requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 45 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by BICR will be reported for participants.
Overall Survival | Up to approximately 59 months
  OS is defined as the time from randomization to death due to any cause. The OS will be reported for all participants.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 45 months
  ORR is defined as the percentage of participants who have a best response of confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 45 months
  DCR is defined, per RECIST 1.1, as the percentage of participants who have achieved Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or demonstrated Stable Disease (SD) for at least 24 weeks. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.) The DCR as assessed by BICR will be presented.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 45 months
  DOR is defined as the time from first documented evidence of CR or PR until the first documented date of disease progression (PD) or death due to any cause, whichever occurs first, for participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 45 months
  PFS is defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS per RECIST 1.1 as assessed by investigator will be reported for participants.
Progression-Free Survival 2 (PFS2) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 45 months
  PFS2 is defined as the time from randomization to subsequent disease progression (PD) per RECIST 1.1 after initiation of a new anticancer therapy, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more lesions and the unequivocal progression of non-target lesions is also considered PD. The PFS2 per RECIST 1.1 as assessed by investigator will be reported for participants.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Change From Baseline in European Organization for Research And Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (GHS) (Item 29) And Quality of Life (QoL) (Item 30) Combined Score | Baseline and up to approximately 25 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change From Baseline in European Organization for Research And Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Functioning (Items 1-5) Combined Score | Baseline and up to approximately 25 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) score will be presented. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (195):
- United States (35):
  - HonorHealth-USOR HonorHealth ( Site 8000), Phoenix, Arizona
  - Moores Cancer Center ( Site 0037), La Jolla, California
  - Kaiser Permanente Riverside Medical Center ( Site 0045), Riverside, California
  - Yale-New Haven Hospital-Smilow Cancer Hospital at Yale-New Haven ( Site 0013), New Haven, Connecticut
  - Mount Sinai Cancer Center ( Site 0018), Miami Beach, Florida
  - Sarasota Memorial Hospital ( Site 0005), Sarasota, Florida
  - Northside Hospital ( Site 0017), Atlanta, Georgia
  - Southeastern Regional Medical Center ( Site 0046), Newnan, Georgia
  - Midwestern Regional Medical Center,Inc. DBA CTCA, Chicago ( Site 0003), Zion, Illinois
  - St. Vincent Hospital and Health Care Center, Inc ( Site 0006), Indianapolis, Indiana
  - Baptist Health Lexington ( Site 0042), Lexington, Kentucky
  - Maryland Oncology Hematology, P.A.-USOR Maryland Oncology Hematology, P.A. ( Site 8002), Rockville, Maryland
  - University of Massachusetts Medical School-Division of Gynecologic Oncology ( Site 0008), Worcester, Massachusetts
  - Karmanos Cancer Institute ( Site 0029), Detroit, Michigan
  - St. Dominic's Hospital ( Site 0024), Jackson, Mississippi
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0026), Hackensack, New Jersey
  - The Blavatnik Family- Chelsea Medical Center at Mount Sinai ( Site 0023), New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone ( Site 0016), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0052), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0009), New York, New York
  - FirstHealth Clinical Trials ( Site 0050), Pinehurst, North Carolina
  - Sanford Medical Center ( Site 0054), Bismarck, North Dakota
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0055), Fargo, North Dakota
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 0039), Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C, Columbus, Ohio
  - Providence Portland Medical Center ( Site 0031), Portland, Oregon
  - Sidney Kimmel Cancer Center - Jefferson Health ( Site 0053), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Magee-Womens Hospital ( Site 0034), Pittsburgh, Pennsylvania
  - AHN West Penn Hospital ( Site 0011), Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion ( Site 0014), Willow Grove, Pennsylvania
  - Sanford Cancer Center-Gynecologic Oncology ( Site 0002), Sioux Falls, South Dakota
  - Texas Oncology - Austin-USOR Texas Oncology - Austin ( Site 8003), Austin, Texas
  - Texas Oncology - Dallas-USOR Texas Oncology - Dallas (Sammons) ( Site 8005), Dallas, Texas
  - Texas Oncology - Tyler-USOR Texas Oncology - Northeast Texas ( Site 8004), Tyler, Texas
  - VCU Health Adult Outpatient Pavillion ( Site 0022), Richmond, Virginia
- Australia (7):
  - Northern Cancer Institute ( Site 0206), St Leonards, New South Wales
  - Westmead Hospital-Department of Gynaecological Oncology ( Site 0201), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Monash Health ( Site 0202), Clayton, Victoria
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0207), Melbourne, Victoria
  - Epworth Freemasons ( Site 0203), Melbourne, Victoria
  - St. John of God Subiaco Hospital-Oncology Clinical Trials Unit ( Site 0204), Subiaco, Western Australia
- Belgium (3):
  - Institut Jules Bordet-Medicine Oncology ( Site 0321), Brussels, Bruxelles-Capitale, Region de
  - Grand Hôpital de Charleroi-Oncology & Hematology ( Site 0323), Charleroi, Hainaut
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman ( Site 0320), Liège, Liege
- Brazil (3):
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 3005), Natal, Rio Grande do Norte
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 3001), São Paulo, São Paulo
  - A. C. Camargo Cancer Center-CAPEC ( Site 3003), São Paulo
- Canada (9):
  - Cross Cancer Institute ( Site 0513), Edmonton, Alberta
  - BC Cancer Kelowna ( Site 0517), Kelowna, British Columbia
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 0518), Vancouver, British Columbia
  - Sunnybrook Health Sciences - Odette Cancer Centre ( Site 0509), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0510), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0519), Montreal, Quebec
  - Jewish General Hospital ( Site 0504), Montreal, Quebec
  - McGill University Health Centre ( Site 0505), Montreal, Quebec
  - Saskatoon Cancer Center-Clinical Research Department ( Site 0520), Saskatoon, Saskatchewan
- Chile (3):
  - FALP-UIDO ( Site 0602), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Centro del Cáncer ( Site 0604), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0603), Santiago, Region M. de Santiago
- China (31):
  - Anhui Provincial Hospital-Obstetrics and Gynecology ( Site 0730), Hefei, Anhui
  - Beijing Obstetric and Gynecology Hospital ( Site 0740), Beijing, Beijing Municipality
  - Peking University First Hospital ( Site 0723), Beijing, Beijing Municipality
  - Beijing Cancer hospital ( Site 0715), Beijing, Beijing Municipality
  - Southwest Hospital of Third Military Medical University ( Site 0719), Chongqing, Chongqing Municipality
  - 2nd Affiliated Hospital Chongqing Medical Universi ( Site 0745), Chongqing, Chongqing Municipality
  - Fuling Central Hospital ( Site 0733), Fulingqu, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0720), Fuzhou, Fujian
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 0710), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College ( Site 0732), Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical College ( Site 0731), Zhanjiang, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital-Gynecological oncology ( Site 0704), Nanning, Guangxi
  - Hainan General Hospital ( Site 0703), Haikou, Hainan
  - Harbin Medical University Cancer Hospital ( Site 0711), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0713), Zhengzhou, Henan
  - Wuhan Union Hospital-Medical Oncology ( Site 0716), Wuhan, Hubei
  - Xiangya Hospital Central South University-Gynecology ( Site 0708), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0709), Changsha, Hunan
  - Jiangsu Province Hospital-Oncology Department ( Site 0707), Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 0729), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 0705), Changchun, Jilin
  - Shaanxi Provincial Cancer Hospital ( Site 0714), Xi'an, Shaanxi
  - Binzhou Medical University Hospital-Oncology department ( Site 0735), Binzhou, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University ( Site 0702), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital-Gynecology department ( Site 0717), Shanghai, Shanghai Municipality
  - West China Second University Hospital Sichuan University ( Site 0701), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 0706), Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital-Gynecology Department ( Site 0721), Kunming, Yunnan
  - The Affiliated Women's Hospital of Zhejiang University-Obstetrics and Gynecology ( Site 0726), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology ( Site 0700), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Gynecology ( Site 0725), Wenzhou, Zhejiang
- Czechia (8):
  - Fakultní nemocnice Brno Bohunice-Gynekologicko-porodnicka klinika ( Site 0404), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Gynekologicko-porodnicka klinika ( Site 0403), Ostrava, Moravskoslezský kraj
  - Nemocnice AGEL Novy Jicin a.s.-Oddeleni radioterapie a onkologie ( Site 0406), Nový Jiín, Novy Jicin
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0402), Olomouc, Olomoucký kraj
  - Vseobecna fakultni nemocnice v Praze-Gynekologicko-porodnicka klinika 1.LF a VFN ( Site 0405), Prague, Praha 2
  - Fakultni nemocnice Bulovka-Gynekologicko-porodnicka klinika ( Site 0401), Prague, Praha 8
  - Nemocnice Tomase Bati ve Zline-Onkologické oddělení ( Site 0407), Zlín, Zlín
  - Fakultni nemocnice Kralovske Vinohrady-Gynekologicko-porodnická klinika ( Site 0408), Prague
- Denmark (4):
  - Rigshospitalet ( Site 0903), Copenhagen, Capital Region
  - Herlev and Gentofte Hospital ( Site 0902), Copenhagen, Capital Region
  - Aalborg Universitetshospital, Syd ( Site 0905), Aalborg, North Denmark
  - Roskilde Sygehus-Oncology department ( Site 0904), Roskilde, Region Sjælland
- Finland (3):
  - Kuopion Yliopistollinen Sairaala ( Site 1002), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala-Gynecology and Obstetrics ( Site 1001), Tampere, Pirkanmaa
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 1003), Helsinki, Uusimaa
- Germany (4):
  - Universitaetsklinikum Ulm ( Site 1106), Ulm, Baden-Wurttemberg
  - Universitätsklinikum Bonn-Gynaecological oncology ( Site 1105), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Frauenheilkunde und Gebur, Dresden, Saxony
  - Charité Campus Virchow-Klinikum ( Site 1103), Berlin
- Országos Onkológiai Intézet-Ngyógyászat ( Site 1201), Budapest, Hungary
- Ireland (2):
  - Bon Secours Cork Hospital ( Site 1305), Cork
  - St. James's Hospital-Cancer clinical trials office ( Site 1301), Dublin
- Israel (5):
  - Soroka Medical Center ( Site 1403), Beersheba
  - Rambam Health Care Campus-Gyneco-oncology unit ( Site 1402), Haifa
  - Edith Wolfson Medical Center-Obstetrics & Gynecology ( Site 1405), Holon
  - Shaare Zedek Medical Center ( Site 1404), Jerusalem
  - Sheba Medical Center ( Site 1401), Ramat Gan
- Italy (10):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Oncologia Sperimentale Uro-Genitale ( Site 1, Napoli, Campania
  - IRCCS - AOU di Bologna-SSD Oncologia medica Addarii ( Site 1503), Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-Oncologia Medica ( Site 1513), Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli-Ginecologia Oncologica ( Site 1502), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Chirurgia Ginecologica ( Site 150, Milan, Lombardy
  - Ospedale Mauriziano-SCDU ONCOLOGIA MEDICA ( Site 1514), Turin, Piedmont
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 1 ( Site 1504), Rome, Roma
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 1509), Florence, Tuscany
  - AULSS8 Berica-Ospedale S.Bortolo-ONCOLOGIA CLINICA ( Site 1510), Vicenza, Veneto
  - Istituto Europeo di Oncologia IRCCS-Divisione di Ginecologia Oncologica ( Site 1506), Milan
- Japan (17):
  - National Cancer Center Hospital East ( Site 1604), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 1611), Matsuyama, Ehime
  - Ehime University Hospital ( Site 1614), Tōon, Ehime
  - Kurume University Hospital ( Site 1612), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center-Gynecology ( Site 1603), Ōta, Gunma
  - Hokkaido University Hospital ( Site 1601), Sapporo, Hokkaido
  - Tsukuba University Hospital ( Site 1618), Tsukuba, Ibaraki
  - Iwate Medical University Hospital ( Site 1602), Shiwa-gun Yahaba-cho, Iwate
  - Niigata University Medical & Dental Hospital ( Site 1613), Chuo-ku, Niigata, Niigata
  - Saitama Medical University International Medical Center ( Site 1605), Hidaka-shi, Saitama
  - Shizuoka Cancer Center ( Site 1609), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 1607), Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research ( Site 1616), Koto, Tokyo
  - The Jikei University Hospital ( Site 1615), Minato-ku, Tokyo
  - Keio university hospital ( Site 1606), Shinjyuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 1608), Fukuoka
  - Osaka International Cancer Institute ( Site 1617), Osaka
- Netherlands (8):
  - Radboudumc-Medical Oncology ( Site 1703), Nijmegen, Gelderland
  - Maastricht UMC+ ( Site 1709), Maastricht, Limburg
  - Catharina Ziekenhuis-Oncology ( Site 1704), Eindhoven, North Brabant
  - Amsterdam UMC, locatie AMC ( Site 1706), Amsterdam, North Holland
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 1702), Leiden, South Holland
  - Erasmus Medisch Centrum-Medical Oncology ( Site 1701), Rotterdam, South Holland
  - University Medical Center Groningen ( Site 1707), Groningen
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 1705), Utrecht
- Auckland City Hospital-Cancer & Blood Research ( Site 1801), Auckland, New Zealand
- Oslo universitetssykehus, Radiumhospitalet ( Site 1901), Oslo, Norway
- Poland (8):
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Me-Oddzial Ginekologii Onkologicznej ( Sit, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej ( Site 2006), Lublin, Lublin Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2007), Siedlce, Masovian Voivodeship
  - Szpital Kliniczny im. Księżnej Anny Mazowieckiej ( Site 2009), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Ginekologii Onkologicznej ( Sit, Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii-Oddzial Onkologii Ginekologicznej ( Site 2003), Bialystok, Podlaskie Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-III Klinika Radioterapii i Chemioterapii ( Site 20, Gliwice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 2010), Kielce, Świętokrzyskie Voivodeship
- Russia (2):
  - Moscow City Oncology Hospital #62 ( Site 2204), Krasnogorsk, Moscow Oblast
  - Yaroslavl Regional Cancer Hospital-Oncology ( Site 2202), Yaroslavl, Yaroslavl Oblast
- South Korea (4):
  - Seoul National University Hospital ( Site 2302), Seoul
  - Severance Hospital, Yonsei University Health System-Gynecologic cancer center ( Site 2301), Seoul
  - Asan Medical Center-Division of Gynecologic Oncology, Dept. of Obstetrics & Gynecology ( Site 2303), Seoul
  - Gangnam Severance Hospital ( Site 2304), Seoul
- Spain (7):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2406), Hospitalet, Barcelona
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 2405), A Coruña, La Coruna
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 2402), Madrid, Madrid, Comunidad de
  - COMPLEJO HOSPITALARIO DE NAVARRA ( Site 2407), Pamplona, Navarre
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 2404), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron ( Site 2403), Barcelona
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 2401), Seville
- Sweden (3):
  - Skånes Universitetssjukhus Lund-Department of Hematology ( Site 2504), Lund, Skåne County
  - Karolinska Universitetssjukhuset Solna ( Site 2502), Solna, Stockholm County
  - Norrlands universitetssjukhus-Cancercentrum ( Site 2503), Umeå, Västerbotten County
- Taiwan (5):
  - Taichung Veterans General Hospital ( Site 2602), Taichung
  - NATIONAL CHENG-KUNG UNI. HOSP. ( Site 2604), Tainan
  - National Taiwan University Hospital ( Site 2603), Taipei
  - Mackay Memorial Hospital ( Site 2601), Taipei
  - Taipei Veterans General Hospital ( Site 2605), Taipei
- Turkey (Türkiye) (6):
  - Istanbul Universitesi Cerrahpasa ( Site 2702), Fatih, Istanbul
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2704), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 2706), Ankara
  - Akdeniz Universitesi Hastanesi ( Site 2701), Antalya
  - Istanbul University Capa Campus-department of obstetrics and gynaecology ( Site 2705), Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma, Istanbul
- United Kingdom (5):
  - St Bartholomew's Hospital ( Site 2804), London, England
  - The Christie ( Site 2807), Manchester, England
  - The Beatson West of Scotland Cancer Centre ( Site 2805), Glasgow, Glasgow City
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 2806), London, London, City of
  - Hammersmith Hospital-Medical Oncology ( Site 2808), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26299&tenant=MT_MSD_9011